CLINICAL TRIAL: NCT03439761
Title: An Open-label Phase I/II Clinical Trial of PT-112 Injection Alone in the Treatment of Patients With Advanced Solid Tumors and Advanced Hepatocellular Carcinoma
Brief Title: An Open-label Phase I/II Clinical Trial of PT-112 Injection for Advanced Solid Tumors and Advanced Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: SciClone Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCI-PT112-ONC-P1-002
Record Dates: First submitted 2018-02-02; First posted 2018-02-20 (Actual); Last update posted 2018-03-16 (Actual); Status verified 2018-03

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Intervention Model Description: PT-112 injection alone-chemotherapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PT-112 Injection (Experimental): PT-112 Injection alone
  Interventions: Drug: PT-112 Injection

INTERVENTIONS:
Drug: PT-112 Injection — PT-112 Injection 28 days constitute a period. The drug is intravenously dripped for 60 minutes at the 1st, 8th and 15th day of each period.

SUMMARY:
Use PT-112 alone for Phase I dose escalation stage: advanced solid tumors, Phase I dose confirmation stage: advanced solid tumors. Phase II hepatocellular carcinoma (HCC). To evaluate the safety and tolerability of PT-112 injection from 250mg/m2 dose level with 3+3 dose escalation design, find Maximum tolerated dose (MTD), Recommended Phase II Dose(RP2D) and evaluate the Pharmacokinetic (PK) profile of PT-112 through Phase I dose escalation stage. Phase I dose confirmation stage: evaluate the safety and tolerability of PT-112 with RP2D, evaluate the anti-tumor effect of PT-112 at RP2D. Phase II stage: evaluate the anti-tumor effect of PT-112 at RP2D in advanced HCC

DETAILED DESCRIPTION:
This is a multicenter, open-label, phase I/II clinical trial that includes the dose escalation stage, dose confirmation stage and phase II stage.

In dose escalation stage, a 3+3 trial design is adopted for dose escalation. Three dose groups are designed: 200, 250 and 300 mg/m2, once weekly; 28 days constitute a period. The drug is intravenously dripped for 60 minutes at the 1st, 8th and 15th day of each period. The safety, tolerability, PK and preliminary antitumor effect of PT-112 injection alone are evaluated. After Dose limited toxicity (DLT) evaluation is completed for all the patients in a dose group, the Safety Monitoring Committee (SMC) will evaluate the safety and PK of the dose group based on the resulting data, and decide whether the dose should be escalated, and whether the dosing regimen or PK sampling points should be adjusted.

After dose escalation is completed, the RP2D is selected by SMC for dose confirmation. Dose confirmation study will include approximately 10 patients each of the following six types of tumors:

Group 1: Hepatocellular carcinoma Group 2: Gastric cancer Group 3: Colorectal cancer Group 4: Non-small cell lung cancer Group 5: Head and neck cancer Group 6: Breast cancer If it is difficult to include the patients with a specific type of tumor, or if the tumor is not sensitive to the efficacy of investigational drug, the SMC may discuss and decide to prematurely terminate inclusion of patients in that group.

After sufficient data are obtained in dose confirmation stage, the SMC may discuss and decide to initiate phase II trial. Phase II trial plans to include about 40 subjects to evaluate the anti-tumor effect and safety of the monotherapy in patients with advanced HCC who have previously received only one systemic anticancer therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old and ≤ 75 years old, male or female
* Local advanced or metastatic solid tumors confirmed by histopathology or cytology that do not respond to standard treatment or have no standard effective treatment (including but not limited to hepatocellular carcinoma, gastric cancer, colorectal cancer, non-small cell lung cancer, head and neck cancer, and breast cancer)
* Compliance with the requirements for type of tumor in the group in dose confirmation stage;
* Eastern Cooperative Oncology Group (ECOG) physical score: 0 or 1
* Lesions that can be assessed by imaging according to the Response evaluation criteria in solid tumors (RECIST) 1.1 (not required in dose escalation stage);
* Expected survival>12 weeks;
* Subjects should have appropriate organ function and should meet the following requirements for laboratory test results before inclusion:

Generally normal bone marrow reserve: absolute neutrophil count (ANC)

≥1.5*10^9/L, platelet count≥100*10^9/L and hemoglobin≥90 g/L; Generally normal liver function: serum albumin ≥3.0 g/dL; bilirubin ≤1.5×upper limits of normal (ULN), Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) ≤ 2.5×ULN, ALT or AST ≤5×ULN for patients with liver metastases or primary liver cancer; Normal renal function: creatinine ≤1.5×ULN or creatinine clearance ≥60ml/min (according to Cockcroft-Gault formula); Generally normal coagulation function: International Normalized Ratio(INR)≤1.5×ULN, activated partial thromboplastin time (APTT) ≤1.5×ULN; Cardiac function: Left ventricular ejection fraction (LVEF)≥ 50%;

* Women of childbearing age (defined as women under 50 years old or above 50 years old who have an amenorrhea period shorter than 12 months before inclusion in the study) who show negative in serum β-human chorionic gonadotrophin (β-HCG) test;
* Subjects with history of brain metastases who are diagnosed with stable disease not requiring treatment with steroid or anticonvulsant, regardless of previous radiotherapy;
* Signing of informed consent form before participation in the study.

Other inclusion criteria for the phase II trial:

* Advanced HCC diagnosed by histopathology or cytology that cannot be surgically removed or progresses after intervention/local treatment, previous treatment with one systemic anti-cancer chemotherapy, Barcelona Clinic Liver Cancer (BCLC) staging: Stage C, Child-Pugh A and mild grade B (≤7);

  * Lesions that can be assessed by imaging according to the RECIST 1.1;

Exclusion Criteria:

* Untreated active hepatitis (hepatitis B: HBsAg positive with abnormal liver function and hepatitis B virus(HBV)-DNA ≥ 2000international unit (IU)/ml; hepatitis C: hepatitis C virus (HCV)-RNA positive and abnormal liver function);
* antitumor immunoregulation therapy, immunosuppressive therapy, corticosteroids > 20 mg/day (unless used to prevent contrast agent reactions during radiotherapy), growth factor therapy (such as erythropoietin) or transfusion therapy within 14 days before use of the investigational drug;
* Unrecovered toxic and side effects caused by previous treatment (CTCAE ≤ grade 1), except hair loss and other tolerable events judged by the investigators;
* Any grade of peripheral neuropathy within 28 days prior to use of the investigational drug;
* Known allergy or hypersensitivity to platinum drugs;
* Antitumor therapy like chemotherapy, biotherapy, radiotherapy, endocrine therapy, target therapy (except Nitrourea, mitomycin C) within 4 weeks before use of the investigational drug. Use Nitrourea or mitomycin C within 6 weeks before use of the investigational drug.
* Major surgery within 28 days before use of the investigational drug;
* Acute bacterial, viral or fungal infections requiring systemic treatment or unexplained fever during screening before the first administration of drug (body temperature> 38.5℃);
* Moderate or massive effusion of body cavity need treatment;
* History of mental illness;
* Human Immunodeficiency Virus(HIV) carriers or Acquired Immune Deficiency Syndrome (AIDS) patients;
* Any of the following conditions within six months before sign informed consent form : uncontrolled congestive heart failure (New York Heart Association grade 2 or 4), angina pectoris, myocardial infarction, stroke (except lacunar infarction), coronary/peripheral artery bypass surgery, pulmonary embolism);
* Uncontrolled arrhythmia or persistent QT interval prolongation, > 450 ms for men or > 470 ms for women;
* Use of any investigational drug or device within 28 days before the use of investigational drug;
* Pregnant or lactating women;
* Women of childbearing age and fertile men who cannot take effective adequate double contraceptives during the study or within three months after completion of the study;
* Any other conditions based on which the investigators believe that the patient should not participate in the study;

Other exclusion criteria for the phase II trial:

* Patients with advanced HCC who have received more than two kinds of systemic chemotherapy (but not including targeted therapies or immunity checkpoint inhibitors like programmed death(PD)-1 or PD-L1 antibody treatment).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2018-03-07 (Actual); Primary Completion 2020-05 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Adverse Event (AE) | Informed consent form (ICF) signed till 28days after end of treatment
  The primary outcome for Phase I dose escalation stage
Dose Limited Toxicity (DLT) | First dose till 28days after 1st dosing. (1st cycle treatment)
  The primary outcome for Phase I dose escalation stage
AE | ICF signed till 28days after end of treatment
  The primary outcome for Phase I dose confirmation stage
Disease Control Rate (DCR) | subject enrolled till disease progress estimate 6 months after first dosing.
  The primary outcome for Phase II (rate of complete response(CR)+partial response (PR)+stable disease(SD))

SECONDARY OUTCOMES:
DCR | subject enrolled till disease progress estimate 6 months after first dosing.
  The secondary outcome for Phase I (rate of CR+PR+SD)
Objective Response Rate (ORR) | subject enrolled till disease progress estimate 6 months after first dosing.
  The secondary outcome for Phase I/II (rate of CR+PR)
Progress Free Survival(PFS) | enrolled study till first disease progress estimate 6 months after first dosing.
  The secondary outcome for Phase I/II
Peak Plasma Concentration （Cmax） | collect PK blood sample in first and second cycles (28 and 56 days after 1st dosing)
  The secondary outcome for Phase I dose escalation stage including: Cmax for PT-112.
Area under the plasma concentration versus time curve (AUC) | collect PK blood sample in first and second cycles (28 and 56 days after 1st dosing)
  The secondary outcome for Phase I dose escalation stage including: AUC for PT-112.
Peak time （Tmax） | collect PK blood sample in first and second cycles (28 and 56 days after 1st dosing)
  The secondary outcome for Phase I dose escalation stage including: Tmax for PT-112
AE | AE from ICF signed till 28days after end of treatment
  The secondary outcome for Phase II

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, MD, Principal Investigator — Shanghai East Hospital
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes